CLINICAL TRIAL: NCT00038883
Title: Campath-1H Snd Allogeneic Blood Stem Cell Transplantation for Lymphoid Malignancies
Brief Title: Campath-1H and Allogeneic Blood Stem Cell Transplantation for Lymphoid Malignancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Leudosite (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-410
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Leukemia, Lymphocytic, Chronic; Leukemia, Lymphocytic, Acute; Lymphoma, Low-Grade; Lymphoma, T-Cell; Lymphoma, B-Cell
Keywords: Lymphoid Malignancies; Chronic Lymphocytic Leukemia; Acute Lymphoblastic Leukemia; Low grade Lymphoma; B and T cell Lymphoma of the intermediate and high grade
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell; Lymphoma, B-Cell | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Campath-1H (Experimental): 10 mg/day x 5
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H — 10 mg/day x 5, starting with the first day of chemotherapy
  Other Names: Alemutuzumab; Campath

SUMMARY:
High dose chemotherapy followed by transplantation of allogeneic hematopoietic stem cell with the use of Campath-1h, a monoclonal antibody that have a synergistic effect to chemotherapy with minimal toxicity. In addition Campath-1H can improve engraftment of donor cells through its immunosuppressive properties.

DETAILED DESCRIPTION:
Alemtuzumab is a drug that is designed to specifically attack some types of leukemia and lymphoma cells. In addition, it weakens the immune system, helping to prevent the rejection of donor marrow or stem cells.

If you are found to be eligible to take part in this study, you will be admitted to the hospital for treatment. Alemtuzumab will be injected into your vein over a period of 4 hours. This will be done 5 days in a row (Days 1 to 5). Drugs diphenhydramine (Benadryl), solumedrol and acetaminophen (Tylenol) will be given in to decrease the risk of or ease side effects before each dose of the alemtuzumab.

You will also receive Carmustine over one hour on the first day. From the second to the fifth day, you will receive cytarabine and etoposide twice a day. On the six day, you will receive melphalan once. Both drugs will be given through a catheter (plastic tube) that extends into the large chest vein. The catheter will be left in place throughout treatment on this study. Some participants, depending on their type of disease, will also receive rituximab. Rituximab will be given during the first day of chemotherapy then once a week for a total of 4 doses.

When chemotherapy is finished, blood stem cells from a donor will be given through the catheter. G-CSF, a growth factor that promotes the production of blood cells, will be injected under the skin once a day until your blood cell counts recover to a certain level.

Blood tests (about 2 tablespoons each) , urine tests, bone marrow aspirations, and x-rays will be done as needed to track the effects of the transplant. The blood tests will be drawn daily while in the hospital and then at least twice weekly as an outpatient for the first 100 days. The CT scans and bone marrow studies will be done at 1, 3, 6, and 12 months and then every 6 months for at least 3 years after transplant. You may also have transfusions of blood and platelets as needed.

You will need to stay in the hospital about 3 to 4 weeks. You will be taken off study if their disease gets worse or intolerable side effects occur. You must stay in the Houston area for about 100 days after the transplant. After that, you will be asked to return to Houston every 6 months for the next 3-5 years for scans (CT, gallium, or PET scans), and bone marrow aspirations over the next 3-5 years.

This is an investigational study. The FDA has approved the drugs used in this study. Their use together in this study is investigational. About 142 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 15-65 years old
2. B or T-cell lymphoid disease, not eligible for non-myeloablative transplantation.
3. Patients in relapse after failing conventional chemotherapy.
4. Patients with HLA-identical or one-antigen mismatched sibling, or a matched unrelated donor.
5. Performance status </=2.

Exclusion Criteria:

1. Past history of anaphylaxis following exposure to rat or mouse derived CDR-grafted humanized monoclonal antibodies.
2. Less than 4 weeks since prior chemotherapy.
3. Pregnancy or lactation.
4. HIV or HTLV-I positivity.
5. Serum creatinine >1.6 mg/dl or serum bilirubin >0.2 mg/dl unless due to tumor, SGPT >/= 2 x NI
6. PFT-DCLO<50%, cardiac EF <50% of predicted levels.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2001-04-09 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
CAMPATH 2-year event-free survival rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org